CLINICAL TRIAL: NCT02833610
Title: A Phase 2, Single-Arm Study of Denosumab in Multiple Myeloma Patients With Renal Insufficiency
Brief Title: A Study of Denosumab in Multiple Myeloma Patients With Renal Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry); Emory University (Other); University of Rochester (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Yee, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-571
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Denosumab Injection (Experimental): Patients will be administered Denosumab Q4W at a pre-determine dose for 12 cycles. Denosumab Q4W is administered by subcutaneous injection.
  Interventions: Drug: Denosumab Q4W

INTERVENTIONS:
Drug: Denosumab Q4W
  Other Names: Xgeva; Prolia

SUMMARY:
This research study is studying a possible therapy as a possible treatment for the consequences of Multiple Myeloma with renal insufficiency.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. This study will assess the safety and tolerability of denosumab in Multiple Myeloma participants, by studying drug interactions with different parts of the body.

The FDA (the U.S. Food and Drug Administration) has not approved Denosumab for this specific disease but it has been approved denosumab for use in other cancers to treat cancer-related bone disease such as prostate and breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic MM as defined by IMWG requiring anti-myeloma therapy.

  * Monoclonal plasma cells in the bone marrow greater than or equal to 10% and/or presence of a biopsy-proven plasmacytoma
  * Monoclonal protein present in the serum and/or urine
* Creatinine clearance < 30 mL/min, not eligible for bisphosphonate. Estimated glomerular filtration rate will be calculated using Cockcroft-Gault equation.
* Serum calcium or albumin-adjusted serum calcium ≥ 2.1 mmol/L (8.4 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL) (Reference range 8.5-10.8 mg/dL)
* Able to tolerate daily supplementation of calcium and vitamin D
* Vitamin D level ≥ 30 ng/mL after repletion
* Participants must have normal organ as defined below:

  * Total bilirubin ≤ 2.0 x ULN
  * AST(SGOT) ≤2.5 × institutional upper limit of normal
  * ALT(SGPT) ≤2.5 × institutional upper limit of normal
* Plan to receive anti-myeloma therapies.
* Age ≥ 18 years.
* ECOG performance status ≤ 2
* Life expectancy greater than 6 months
* 0-3 lines of prior anti-myeloma therapy.
* Subjects with reproductive potential must be willing to use, in combination with his/her partner, 2 highly effective methods of effective contraception or practice sexual abstinence throughout the study and continue for 5 months after the study duration. Subjects who are surgically sterile (e.g. history of bilateral tubal ligation, hysterectomy) or whose sexual partner is sterile (e.g. history of vasectomy) are not required to use additional contraceptive measures.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior administration of denosumab.
* Active IV bisphosphonate use in the last 3 months.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Plasma cell leukemia.
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw.
* Active dental or jaw condition which requires oral surgery, including tooth extraction.
* Non-healed dental/oral surgery, including tooth extraction.
* Planned invasive dental procedures during the course of study.
* Evidence of any of the following conditions per subject self-report or medical chart review

  * Any prior invasive malignancy within 5 years of enrollment that may affect outcome of study
  * Any non-invasive malignancy not treated with curative intent or with known active disease within 5 years before enrollment that may affect outcome of study
  * Major surgery or significant traumatic injury occurring within 4 weeks before enrollment
  * Active infection with Hepatitis B virus or Hepatitis C virus
  * known infection with human immunodeficiency virus (HIV)
  * Active infection requiring IV anti-infective therapy
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 months after the end of treatment.
* Female subject of child-bearing potential is not willing to use, in combination with her partner, 2 methods of highly effective contraception during treatment and for 5 months after the end of treatment.
* Clinically significant hypersensitivity to denosumab 120 mg.
* Known sensitivity to any of the products to be administered during the study (e.g. calcium, or vitamin D).
* Subject is receiving or is less than 14 days since ending other experimental drug (no marketing authorization for any indication).
* Any major medical or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Percent Change Of sCTX Levels | 2 years

SECONDARY OUTCOMES:
Percent Change In Bone Mineral Density | 2 years
Percent Change In uNTX Levels | 2 years
Subject Incidence Of Hypocalcemia | 2 years
Subject Incidence Of Occurrence Of Documented SRE At 12 Months | 2 years
Subject Incidence Of Adverse Events | 2 years
Percent Change In Bone Turnover Markers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth K O'Donnell, MD, Principal Investigator — Massachusetts General Hospital
Locations (7):
- United States (7):
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Newton Wellesley Hospital, Newton, Massachusetts
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No